CLINICAL TRIAL: NCT03143192
Title: Treatment of Diabetic Macular Edema With Aflibercept and Micropulse Laser
Acronym: DAM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Keyvan Koushan (Other)
Responsible Party: Sponsor-Investigator, Keyvan Koushan, Principal Investigator, Toronto Retina Institute
Organization: Toronto Retina Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19228
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Macular Edema
Keywords: DME, Micropulse Laser, Anti-VEGF

STUDY DESIGN:
Intervention Model Description: This will be a parallel study comparing the results of patients who receive aflibercept and micropulse laser versus those who only receive aflibercept. The second group will receive sham laser to prevent placebo effects.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and technicians (measuring ocular coherence tomography, fluorescein auto fluorescence and visual acuity) will be masked. The investigator and study coordinator will be unmasked to direct the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept with Micropulse Laser (Experimental): Aflibercept 2mg (0.05mL) injected intravitreally every 4 weeks or as needed Micropulse Laser at initial visit and reassessed every 12 weeks.
  Interventions: Combination Product: Micropulse Laser
- Aflibercept with Sham Laser (Sham Comparator): Aflibercept 2mg (0.05mL) injected intravitreally every 4 weeks or as needed Sham Laser at initial visit and reassessed every 12 weeks.
  Interventions: Device: Sham Laser

INTERVENTIONS:
Combination Product: Micropulse Laser — Aflibercept injection with Micropulse laser.
  Arms: Aflibercept with Micropulse Laser
Device: Sham Laser — Aflibercept injection with Sham Laser
  Arms: Aflibercept with Sham Laser

SUMMARY:
The goal of this pilot study is to investigate the safety and efficacy of micropulse (MP) macular laser in combination with intravitreal aflibercept for the treatment of centre-involved diabetic macular edema.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is one of the major causes of visual decline among diabetic patients. Early Treatment of Diabetic Retinopathy Study has established focal/grid macular laser as the standard of treatment for clinically significant macular edema. More recently, intravitreal injections of anti-VEGF agents, either as monotherapy or in combination with focal/grid laser, have proven to be superior for the treatment of DME compared to laser alone.

Micropulse (MP) macular laser involves applying the laser in a fraction of the time within very small pockets of energy. Unline traditional focal/grid macular laser, the micropulse method of delivery does not leave any visible burns on the retina.

A recent release by the Diabetic Retinopathy Clinical Research Network has shown that deferring focal/grid laser and treating diabetic macular edema with only anti-VEGF may lead to better visual outcomes. Since MP laser does not have the undesired side effect of leaving laser scars on the macula, the study is to show that prompt MP laser in addition to anti-vegf injections may lead to better visual outcomes and/or decreased treatment burden without the undesired side effect of macular scarring.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II Diabetes Mellitus
* Presence of centre-involved Diabetic Macular Edema (DME) with the Central Macular Thickness (CMT) of ≥ 310µm on the spectral-domain Optical Coherence Tomography (OCT)
* Best corrected Visual Acuity (BCVA) between, and including, 20/30 and 20/400 in the study eye.
* Patient's willingness and ability to attend the study visits

Exclusion Criteria:

* Any other potential causes of macular edema such as active uveitis, epiretinal membrane, post-operative CME, and vitromacular traction
* Any history of major intraocular surgery (such as cataract surgery or vitrectomy) in the study eye within prior six months, or anticipated need for intraocular surgery within the next six months from the enrollment
* Any major ocular pathology limiting potential vision such as large macular scars, vitreous hemorrhage, corneal opacities, visually significant cataracts, advanced glaucoma, or other types of optic neuropathy
* Any history of Panretinal Photocoagulation (PRP) in the study eye or anticipated need for PRP within the next 6 months from enrollment
* Any history of DME treatment (focal laser, anti-VEGF, or intraocular/periocular steroids) in the study eye in the past 4 months prior to the enrollment
* Significant renal disease requiring dialysis
* Significant heart disease, stroke or transient ischemic attack requiring hospitalization in the past 4 months prior to the study
* Presence of active ocular or periocular infection
* Presence of active intraocular inflammation
* Known hypersensitivity to aflibercept or to any ingredient in the formulation or to any component of the container

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Number of injections for each group | 48 weeks
  Number of intravitreal injections for each group

SECONDARY OUTCOMES:
Changes in visual acuity | 24 weeks
  Changes in visual acuity from baseline to 24 adjusted for baseline
Changes in visual acuity | 48 weeks
  Changes in visual acuity from baseline to 48 weeks adjusted for baseline
Changes in OCT Central Macular Thickness and Volume | 24 weeks
  Measurement changes in central macular thickness at 24 weeks
Changes in OCT Central Macular Thickness and Volume | 48 weeks
  Measurement changes in central macular thickness at 48 weeks
Number of injections half way | 24 weeks
  Number of intravitreal injections of each group at 24 weeks
Proportion of eyes with 2 or 3 lines of visual gain or loss | 24 weeks
  Improvement or deterioration of vision of 2 or 3 lines at 24 weeks
Proportion of eyes with 2 or 3 lines of visual gain or loss | 48 weeks
  Improvement or deterioration of vision of 2 or 3 lines at 48 weeks
Proportion of eyes that achieve 20/20 vision | 24 weeks
  Eyes that are able to see 20/20 at 24 weeks regardless of baseline
Proportion of eyes that achieve 20/20 vision | 48 weeks
  Eyes that are able to see 20/20 at 48 weeks regardless of baseline
Proportion of eyes that have PRP, vitreous hemorrhage, and vitrectomy. | 48 weeks
  Proportion of eyes in each study group that require panretinal photocoagulation, have a vitreous hemorrhage, or require a vitrectomy during the course of the study.
Proportion of eyes that had vision or OCT improvement | 48 weeks
  In patients with HbA1c ≤ 8% or separately measured in patients with HbA1C > 8%

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Koushan, MD, FRCSC, Principal Investigator — Toronto Retina Institute
Locations (2):
- Canada (2):
  - Mississauga Retina Institute, Mississauga, Ontario
  - Toronto Retina Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
The results of this study will be analyzed statistically which will be shared with other members of the scientific community but the individual participant data along with their identifiers will not be available to other researchers.

REFERENCES:
- [Derived] Koushan K, Eshtiaghi A, Fung P, Berger AR, Chow DR. Treatment of Diabetic Macular Edema with Aflibercept and Micropulse Laser (DAM Study). Clin Ophthalmol. 2022 Apr 8;16:1109-1115. doi: 10.2147/OPTH.S360869. eCollection 2022. PMID 35422607